CLINICAL TRIAL: NCT05656027
Title: A Multi-Center, Double-Masked Phase 3 Evaluation of the Safety and Efficacy of LNZ101 for the Treatment of Presbyopia
Brief Title: Phase 3 Evaluation of the Safety and Efficacy of LNZ101 for the Treatment of Presbyopia
Acronym: CLARITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-150-0015
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia; Refractive Error; Near Vision; Miosis; Eye Diseases
Keywords: Pharmaceutical Solutions; Eye Drops; CLARITY; Presbyopia; Ophthalmic Solutions; Miotic
MeSH Terms: conditions — Presbyopia; Refractive Errors; Myopia; Miosis; Eye Diseases | interventions — aceclidine; Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: A multi-center, double-masked, randomized, active-controlled, safety and efficacy study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aceclidine + Brimonidine (LNZ101) dosed bilaterally (Experimental): LNZ101 (Aceclidine /Brimonidine) ophthalmic solution
  Interventions: Drug: Aceclidine + Brimonidine
- Aceclidine Ophthalmic Solution (LNZ100) dosed bilaterally (Experimental): LNZ100 (Aceclidine) ophthalmic solution
  Interventions: Drug: Aceclidine
- Brimonidine ophthalmic solution dosed bilaterally (Experimental): Brimonidine ophthalmic solution
  Interventions: Drug: Brimonidine

INTERVENTIONS:
Drug: Aceclidine + Brimonidine — LNZ101 (Aceclidine/Brimonidine) ophthalmic solution
  Arms: Aceclidine + Brimonidine (LNZ101) dosed bilaterally
Drug: Aceclidine — LNZ100 Aceclidine ophthalmic solution
  Arms: Aceclidine Ophthalmic Solution (LNZ100) dosed bilaterally
Drug: Brimonidine — Brimonidine ophthalmic solution
  Arms: Brimonidine ophthalmic solution dosed bilaterally

SUMMARY:
Phase 3 study to evaluate the safety and effectiveness of LNZ101 for the treatment of Presbyopia.

DETAILED DESCRIPTION:
Phase 3 study to evaluate the safety and effectiveness of LNZ101 compared with LNZ100 and Brimonidine for the treatment of Presbyopia.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent and sign a Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed;
2. Be able and willing to follow all instructions and attend all study visits;
3. Be 45-75 years of age of either sex and any race or ethnicity at Visit 1;
4. Have +1.00 to -4.00 diopter (D) of sphere calculated in minus cylinder (so that spherical equivalent (SE) results in myopia no more severe than -4.00 D MRSE) in both eyes determined by manifest refraction documented at Visit 1;
5. Have ≤2.00 D of cylinder (minus cylinder) in both eyes determined by manifest refraction documented at Visit 1;
6. Be presbyopic as determined at Visit 1

Exclusion Criteria:

Subjects must not:

1. Be a female of childbearing potential who is currently pregnant, nursing, or planning a pregnancy;
2. Have known contraindications or sensitivity to the use of any of the study medications or their components;
3. Have an active ocular infection at Visit 1 or at Visit 2 (bacterial, viral, or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation in either eye;
4. Have moderate or severe dry eye defined as total central corneal fluorescein staining in either eye at Visit 1;
5. Have clinically significant abnormal lens findings including early lens changes in either eye during dilated slit-lamp biomicroscopy and fundus exam documented within 3 months of Visit 1 or at Visit 1;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 3 hours post-treatment in the study eye
  Efficacy Study of the percentage of subjects who achieve a 3-line or greater improvement from baseline in the study eye with no loss in BCDVA ≥ 5 letters (ETDRS chart at 4 m).

CONTACTS AND LOCATIONS:
Overall Officials: Alisyn Facemire, BA, Study Director — LENZ Therapeutics
Locations (20):
- United States (20):
  - Site #106, Chandler, Arizona
  - Site #121, Mesa, Arizona
  - Site #122, Phoenix, Arizona
  - Site #124, Phoenix, Arizona
  - Site #125, Sun City, Arizona
  - Site #110, Garden Grove, California
  - Site #101, Glendale, California
  - Site #107, Petaluma, California
  - Site #126, Rancho Cordova, California
  - Site #111, Santa Barbara, California
  - Site #109, Littleton, Colorado
  - Site #102, Mt. Dora, Florida
  - Site #118, Rock Island, Illinois
  - Site #108, Pittsburg, Kansas
  - Site #104, Fargo, North Dakota
  - Site #103, Kingston, Pennsylvania
  - Site #116, Memphis, Tennessee
  - Site #112, Smyrna, Tennessee
  - Site #119, San Antonio, Texas
  - Site #123, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No